CLINICAL TRIAL: NCT03928678
Title: Enhanced Recovery After Surgery Program (ERAS) in Colorectal Cancer Surgery
Brief Title: Implementation of Enhanced Recovery After Surgery Program (ERAS) in Colorectal Cancer Surgery, a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 458
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2020-04

CONDITIONS: Cancer of Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thefast track (FTS group) (Active Comparator)
  Interventions: Procedure: enhanced recovery after surgery program in colorectal cancer surgery
- Thecontrolgroup (Placebo Comparator)
  Interventions: Procedure: enhanced recovery after surgery program in colorectal cancer surgery

INTERVENTIONS:
Procedure: enhanced recovery after surgery program in colorectal cancer surgery — to determine the feasibility of implementation of the ERAS protocol in our institute and its impact on hospital length of stay and outcome of surgery.

SUMMARY:
The aim of our study is to determine the effect of implementation of the ERAS (enhanced recovery after surgery) protocol in our institute and its impact on hospital length of stay and outcome of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 60 years,
* Good nutrition,
* No systemic infection and
* Elective laparoscopic surgery

Exclusion Criteria:

* Age >75 years,
* Malnutrition or an organ system infection
* Associated with obstruction, bleeding, emergency surgery or other surgical intervention
* Tumor with extensive metastasis
* Prior to surgery, patient was fasting, underwent gastrointestinal decompression and received nutritional support
* Previous history of abdominal surgery
* Patient have previously undergone gastrostomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
length of hospital stay in days | 4 days
  length of hospital stay in days

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided